CLINICAL TRIAL: NCT03549104
Title: A Cognitive Behavioral Intervention to Reduce Fear of Hypoglycemia in Young Adults With T1DM
Brief Title: A Cognitive Behavioral Therapy (CBT) Intervention to Reduce Fear of Hypoglycemia in Type 1 Diabetes
Acronym: CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Loyola University Chicago (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Pamela Martyn-Nemeth, Assistant Professor Biobehavioral Nursing Science College of Nursing, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-0382; R21DK116146 (NIH)
Record Dates: First submitted 2018-04-24; First posted 2018-06-07 (Actual); Results first posted 2022-05-20 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: fear of hypoglycemia; glycemic control; glycemic variability; self-management behavior
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal Investigator and outcome assessors masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fear Reduction Efficacy Evaluation (FREE) (Experimental): The FREE intervention group will participate in eight weekly individual one-hour sessions using CBT and exposure treatment for specific fears.
  Interventions: Behavioral: Fear Reduction Intervention
- Attention Control (Active Comparator): The attention control group will participate in eight weekly individual one-hour Diabetes Self-Management Education (DSME) sessions.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Fear Reduction Intervention — FREE
  Arms: Fear Reduction Efficacy Evaluation (FREE)
Behavioral: Attention Control — DSMES
  Arms: Attention Control

SUMMARY:
All persons with type 1 diabetes are at risk for developing hypoglycemia (low blood sugar). This is a life-threatening condition that leads to profound fear of hypoglycemia and reduced quality of life. Fear of hypoglycemia results in glucose fluctuations (from high to low glucose levels). Young adults are particularly at risk because they report high levels of fear of hypoglycemia and poor glucose control. Currently, no diabetes self-management programs specifically address how to cope with fear of hypoglycemia. The investigators propose to pilot test a fear reduction intervention (Fear Reduction Efficacy Evaluation [FREE]) and its effects on fear of hypoglycemia, diabetes self-management, glucose control, and glucose variability.

DETAILED DESCRIPTION:
In persons with type 1 diabetes (T1DM), hypoglycemia is the major limiting factor in achieving optimal blood glycemic control. All persons with T1DM are at risk for hypoglycemia (blood glucose level < 70 mg/dl), which is life-threatening and accompanied by serious physical and psychological symptoms, resulting in a profound fear of hypoglycemia (FOH) and reduced quality of life. Young adults with T1DM are at greater risk for FOH and have worse glycemic control and self-management behavior than other age groups with T1DM. The investigator's preliminary research identified that 77% of young adults with T1DM reported FOH, and FOH resulted in increased glycemic variability. Glycemic variability (GV) is the minute-to-minute fluctuation in blood glucose that can be missed if looking only at A1C, a longer-term measure. Increased GV is dangerous because it is associated with cardiovascular events and diabetes complications. A major gap exists in how to manage FOH as a component of diabetes self-management. The Investigators specifically aim to: (1) determine the feasibility and acceptability of a fear reduction program in young adults with T1DM, who experience FOH; and (2) determine the impact of an 8-week cognitive behavioral therapy (CBT)-based intervention on the outcomes: FOH, self-management behavior, glycemic control, and GV. To achieve these aims, the investigators propose a randomized controlled trial in 50 young adults aged 18 to 35 years with T1DM. At completion, FOH will be measured and glycemic patterns will be analyzed to determine differences between the FREE and control groups. Findings from this proposed pilot study will serve as the foundation for a larger clinical trial to reduce FOH and improve self-management, glycemic control, and GV. This program of research promises to reduce the development of diabetes complications and improve quality of life for young adults with T1DM.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of T1DM ≥ 1 year, receive medical care from an endocrinologist, use insulin pump therapy or multiple daily injection (MDI), have fear of hypoglycemia (screening questionnaire), and attended a basic diabetes educational program

Exclusion Criteria:

Pregnant or breastfeeding, have received therapy specifically for fear of hypoglycemia, have a co-existing chronic illness

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Martyn-Nemeth, PhD, Principal Investigator — University of Illinois at Chic
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martyn-Nemeth P, Duffecy J, Quinn L, Park C, Reutrakul S, Mihailescu D, Park M, Penckofer S. FREE: A randomized controlled feasibility trial of a cognitive behavioral therapy and technology-assisted intervention to reduce fear of hypoglycemia in young adults with type 1 diabetes. J Psychosom Res. 2024 Jun;181:111679. doi: 10.1016/j.jpsychores.2024.111679. Epub 2024 Apr 20. PMID 38677235
- [Derived] Martyn-Nemeth P, Duffecy J, Quinn L, Park C, Mihailescu D, Penckofer S. A cognitive behavioral therapy intervention to reduce fear of hypoglycemia in young adults with type 1 diabetes (FREE): study protocol for a randomized controlled trial. Trials. 2019 Dec 30;20(1):796. doi: 10.1186/s13063-019-3876-4. PMID 31888691

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was administratively removed immediately following consent and randomization. Specifically, 4 hours later, we were contacted by the participant because they had developed a situation (unrelated to the study) that rendered them ineligible to participate.
Period: Overall Study
Arm/Group | Fear Reduction Efficacy Evaluation (FREE) | Attention Control
Started | 25 | 25
Completed | 19 | 21
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Covid shelter in place | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fear Reduction Efficacy Evaluation (FREE) | Attention Control | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (5.5) | 26.1 (4.8) | 26.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 22 | 18 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 21 | 18 | 39
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Fear of hypoglycemia [Mean (Standard Deviation); unit: units on a scale] — Hypoglycemia Fear Scale II - Worry Subscale
  units on a scale | 36.3 (11.8) | 40.7 (11.4) | 38.6 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Fear of Hypoglycemia
Description: Change in Worry Subscale score. Fear of hypoglycemia is measured with the Worry Subscale of the Hypoglycemia Fear Survey II (HFS-II) which is an 18-item, 5-point Likert-style scale with a possible score range from 0-72. A higher score indicates greater fear of hypoglycemia.
Time Frame: Assessing change between two time points: from baseline to week 8 of intervention.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Fear Reduction Efficacy Evaluation (FREE) | Attention Control
Number analyzed (Participants) | 19 | 21
units on a scale
  Week 0 | 54.3 (2.4) | 58.7 (2.3)
  Week 8 | 35.29 (1.7) | 49.0 (2.7)
Statistical Analysis 1: Comparison: Fear Reduction Efficacy Evaluation (FREE) vs Attention Control; Test type: Other; We will evaluate the effects of within-group and between-group differences from baseline (Week 0) to program completion (Week 8) to calculate effect sizes for sample size estimation for a future larger study

2. Secondary Outcome: Glycemic Control
Description: Change in HemoglobinA1c (A1C)
Time Frame: Assessing change between two time points: from baseline to week 8 of intervention.
Measure: Mean (Standard Error); unit: percentage of HbA1C
Arm/Group | Fear Reduction Efficacy Evaluation (FREE) | Attention Control
Number analyzed (Participants) | 18 | 21
percentage of HbA1C
  Week 0 | 7.25 (0.29) | 7.07 (0.19)
  Week 8 | 6.68 (.26) | 6.69 (.20)
Statistical Analysis 1: Comparison: Fear Reduction Efficacy Evaluation (FREE) vs Attention Control; Test type: Other; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Glycemic Variability
Description: Change in glucose variability (continuous glucose monitor-derived, glucose (mg/dl) standard deviation. Higher numbers indicate worse glycemic variability.
Time Frame: Assessing change between two time points: from baseline to week 8 of intervention
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Fear Reduction Efficacy Evaluation (FREE) | Attention Control
Number analyzed (Participants) | 18 | 21
mg/dL
  Week 0 | 57.8 (3.54) | 56.2 (2.7)
  Week 8 | 54.9 (3.4) | 55.5 (3.8)
Statistical Analysis 1: Comparison: Fear Reduction Efficacy Evaluation (FREE) vs Attention Control; Test type: Other; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: Definitions do not differ
Arm/Group | Fear Reduction Efficacy Evaluation (FREE) | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03549104/Prot_SAP_000.pdf